CLINICAL TRIAL: NCT03299647
Title: Effects of Polyunsaturated Fatty Acids on the Visual Memory of Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201705134RINC
Record Dates: First submitted 2017-09-25; First posted 2017-10-03 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: Attention-deficit/hyperactivity disorder; behavioral deficits; cognitive function; polyunsaturated fatty acids; visual memory
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The biospecimen includes plasma and DNA of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD group: Subjects with clinical diagnosis of ADHD according to the DSM-V criteria
- TD group: Typically development controls without lifetime diagnosis with ADHD

SUMMARY:
The investigators anticipate to identify specific polyunsaturated fatty acids that show significant differences between ADHD and control groups. In addition, these findings may offer more biological understanding in explaining the relationship between polyunsaturated fatty acids and visual memory among children with ADHD. The results will significantly contribute to the knowledge of the pathophysiological mechanisms of ADHD, especially the polyunsaturated fatty acids related to the behavioral/visual memory deficits of ADHD.

DETAILED DESCRIPTION:
Because attention deficit hyperactivity disorder (ADHD) is an early onset and long-term impairing disorder with tremendous impact on individuals, families, and societies, detection and diagnosis are very important for ADHD. According to the investigators' previous work, children with ADHD have visual memory deficits as well as inattentive deficits. Previous studies show that polyunsaturated fatty acids are associated with cognitive problems in children. Analyzing differences in polyunsaturated fatty acids between children with ADHD and healthy controls could provide insight into underlying disease pathology of cognitive deficits. In this one-year project, the researchers will perform an analysis of polyunsaturated fatty acids in serum to identify potential biomarkers for the visual memory deficits of ADHD.

The purpose of this study is to:

1. To identify the specific polyunsaturated fatty acids of ADHD symptoms;
2. To identify the relationship between specific polyunsaturated fatty acids and visual memory deficits of ADHD.

This is a one-year project. After careful calculation of sample size, the study will recruit 35 children with ADHD, aged 7-18, and 35 healthy controls with matched age, sex and BMI. The investigators will quantify the polyunsaturated fatty acids in serum. The behavioral measures include ADHDRS-IV, SNAP-IV, CBCL, CGI-ADHD-S, SAICA, and Family APGAR-C. The Cambridge Neuropsychological Test Automated Battery (CANTAB) will be used to assess the visual memory of all participants. Conditional logistic regression and partial least squares discriminant analysis will be applied to identify significant polyunsaturated fatty acids for ADHD and visual memory deficits.

ELIGIBILITY:
Inclusion Criteria:

Patients with ADHD are eligible to be included in this study only if they meet all of the following criteria:

1. Patients will be outpatients who are between 7 and 18 years of age.
2. Patients must have ADHD that meet the Diagnostic and Statistical Manual of Mental disorders, 5th edition (DSM-V) disease diagnostic criteria assessed by the investigator's clinical evaluation, as well as confirmed by the Chinese version of the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Epidemiological Version (K-SADS-E).
3. Patients must have a Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) score > 4 at baseline.
4. Patients must be psychotropic drug-naïve. Patients will be considered to be drug-naïve if they have never received medications specifically to treat ADHD.
5. Patients and parents (or legal representative) must have a degree of understanding sufficient to be able to communicate suitably with the investigator.
6. Patients must be of normal intelligence in the judgment of the investigator. Normal intelligence is defined as achieving a score of 80 or more when IQ testing is administrated.
7. Patients must have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests, including neuropsychological testing and venipunctures.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Patients with current or past history of schizophrenia, schizoaffective Disorder, organic psychosis, bipolar I or II disorder, autism, or autism spectrum disorder. Other comorbid psychiatric disorders are not excluded if the ADHD symptoms are the primary source of impairment for the patient.
2. Patients with a history of any seizure disorder (other than febrile convulsion) or patients who are taking anticonvulsants for seizure control.
3. Patients have been at serious suicidal risk, determined by the investigator.
4. Patients with a history of alcohol or drug abuse within the past 3 months, or who are currently using alcohol, drugs of abuse, or any described or over-the-counter medication in a manner that the investigator considers indicative of abuse.
5. Patients with cardiovascular disease or other conditions that could be aggravated by an increased heart rate or increased blood pressure.
6. Patients who are likely to need Chinese medicine or health-food supplements that have central nervous system activity.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The researchers plan to recruit 35 ADHD subjects and 35 control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Psychiatric interview | 1 hour
  Subjects will be interviewed by Chinese Version of the Kiddie Epidemiologic version of the Schedule for Affective Disorders and Schizophrenia (K-SADS-E)

SECONDARY OUTCOMES:
Continuous Performance Test (CPT) | 15 minutes
  The main feature of CPT is that a rapid presentation of visual or auditory stimuli over a definite period of time. The subjects respond by pressing a switch button in response to a critical stimulus.
Wechsler Intelligence Scale for Children-3rd edition (WISC-III) | 1.5 hours
  The WISC-III is composed of 13 subtests to test children's cognitive ability of different dimensions, which are grouped into two scores: performance IQ score (7 subtests: Picture Completion, Block Design, Object Assembly, Picture Arrangement, Coding, Symbol Search and Mazes subtests) and verbal IQ score (Information, Comprehension, Arithmetic, Similarities, Digit Span and Vocabulary subtests) (Allen and Thorndike 1995).
Cambridge Neuropsychological Test Automated Batteries (CANTAB) | 1.5 hours
  The CANTAB is a computer-administered, nonverbal (visually-presented) set of neuropsychological tasks developed at the University of Cambridge.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yung Shang, MD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No